CLINICAL TRIAL: NCT02400138
Title: Effects of Home-based Respiratory Training After Stroke: A Randomized Controlled Trial
Brief Title: Home-based Respiratory Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Luci Fuscaldi Teixeira-Salmela, Titular professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTS-01
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory training (Experimental): Respiratory training will include training of the inspiratory and expiratory muscles seven times per week over eight weeks, during 40 minutes per day, divided into two 20-min sessions (morning and afternoon). Each 20-min session comprised 4-min sets of respiratory training, followed by 1-min rest between the sets. The training program will be carried-out with the Orygen Dual Valve device, regulated at 50% of the subjects' maximal inspiratory and expiratory pressure values. Once a week, the treating physiotherapist performed a home visit, measured the current values of inspiratory and expiratory strength, and progressed the load to 50% of the new values.
  Interventions: Other: Respiratory training
- Control (Sham Comparator): The control/sham group will underwent exactly the same protocol and weekly monitoring at home, but the participants will receive the devices without resistance of the spring, which will be also concealed. The control group will also attend the weekly sessions and undergo the same procedures, except for the load adjustments. If the training proves to be effective, the control subjects will be informed and have the choice to receive the training with proper loads.
  Interventions: Other: Control

INTERVENTIONS:
Other: Respiratory training — Respiratory training will include training of the inspiratory and expiratory muscle seven times per week over eight weeks, during 40 minutes, divided into two 20-min sessions (morning and afternoon). Each 20-min session comprised 4-min sets of respiratory training, followed by 1-min rest between the sets. The training program will be carried-out with the Orygen Dual Valve regulated at 50% of the subjects' maximal inspiratory and expiratory pressure values. Once a week, the treating physiotherapist performed a home visit, measured the current values of inspiratory and expiratory strength, and progressed the load to 50% of the new values.
  Arms: Respiratory training
Other: Control — The control/sham group will underwent exactly the same protocol and weekly monitoring at home, but the participants will receive the devices without resistance of the spring.
  Arms: Control

SUMMARY:
Weakness of the respiratory muscles demonstrated by individuals with stroke, may generate important symptoms, such as fatigue and dyspnea. Since adequate strength of the inspiratory and expiratory muscles is required, mainly when performing physical activities, rehabilitation interventions for stroke subjects should include respiratory training. This study will test the hypothesis that home-based combined training of the inspiratory and expiratory muscles is effective in improving strength of the inspiratory and expiratory muscles, endurance of the inspiratory muscles, dyspnea, walking capacity, and ocurrence of respiratory complications after stroke. For this clinical trial, people after stroke will be randomly allocated into either experimental or control/sham groups. The experimental group will undertake training of the inspiratory plus expiratory muscles with the Orygen Dual Valve device, regulated at 50% of the subjects' maximal inspiratory and expíratory pressure values, seven times/week over eight weeks during 40 minutes/day. The control group will undertake the same protocol, but the participants will receive the devices without resistance. At baseline, post intervention, and four weeks after the cessation of the intervention, researchers blinded to group allocations will collect the following outcome measures: maximal inspiratory and expiratory pressures, inspiratory endurance, dyspnea, walking capacity, and ocurrence of respiratory complications.

DETAILED DESCRIPTION:
Rationale: Weakness of the respiratory muscles demonstrated by individuals with stroke, may generate important symptoms, such as fatigue and dyspnea. Since adequate strength of the inspiratory and expiratory muscles is required, mainly when performing physical activities, rehabilitation interventions for stroke subjects should include respiratory training.

Aim: This study will test the hypothesis that home-based combined inspiratory muscular training (IMT) plus expiratory muscular training (EMT) program is effective in improving strength of the inspiratory and expiratory muscles, endurance of the inspiratory muscles, dyspnea, walking capacity, and ocurrence of respiratory complications after stroke.

Design: For this prospective, double-blinded, randomized clinical trial, people after stroke will be randomly allocated into either experimental or control/sham groups. The experimental group will undertake training of the inspiratory plus expiratory muscles with the Orygen Dual Valve, regulated at 50% of the subjects' maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) values, seven times/week over eight weeks during 40 minutes/day. The control group will undertake the same protocol, but the participants will receive the devices without resistance. At baseline, post intervention, and four weeks after the cessation of the intervention, researchers blinded to group allocations will collect all outcome measures.

Study outcomes: Primary outcomes will be MIP. Secondary outcomes will include MEP, inspiratory endurance, dyspnea, walking capacity, and ocurrence of respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

Stroke survivors will be eligible if they: were >3 months and <5 years after their last episode of stroke; were >20 years of age; their maximal inspiratory pressure was <80 cmH2O or maximal expiratory pressure was <90 cmH2O [18]; were not undertaking any respiratory training; and were able to provide informed consent.

Exclusion Criteria:

Subjects will be excluded if they had cognitive deficits, facial palsy, associated respiratory diseases, or unstable conditions which might prevent measurement or training; or undergone thoracic or abdominal surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | Baseline (week 0), after training (week 8) and one-month follow-up (weeks 12)
  Changes in maximal inspiratory pressures will be assessed by a digital manovacuometer, following previously described protocols.

SECONDARY OUTCOMES:
Maximal expiratory pressure | Baseline (week 0), after training (week 8) and one-month follow-up (weeks 12)
  Changes in maximal expiratory pressures will be assessed by a digital manovacuometer, following previously described protocols.
Inspiratory endurance | Baseline (week 0), after training (week 8) and one-month follow-up (weeks 12)
  Changes in inspiratory endurance will be assessed by the powerbreathe device, following previously described protocols.
Dyspnea | Baseline (week 0), after training (week 8) and one-month follow-up (weeks 12)
  Changes in dyspnea will be assessed by the Medical Research Council Scale.
Ocurrence of respiratory complications | Baseline (week 0), after training (week 8) and one-month follow-up (weeks 12)
  Changes in ocurrence of respiratory complications will be assessed by asking the participants, whether and how often they were admitted to a hospital, due to respiratory reasons.
Walking capacity | Baseline (week 0), after training (week 8) and one-month follow-up (weeks 12)
  Changes in walking capacity will be evaluated by the six-minute walking test

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Rodrigues-de-Paula, Ph.D., Study Director — Federal University of Minas Gerais
Locations (2):
- Brazil (2):
  - Department of Physical Therapy, Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - NeuroGroup Laboratory, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sutbeyaz ST, Koseoglu F, Inan L, Coskun O. Respiratory muscle training improves cardiopulmonary function and exercise tolerance in subjects with subacute stroke: a randomized controlled trial. Clin Rehabil. 2010 Mar;24(3):240-50. doi: 10.1177/0269215509358932. Epub 2010 Feb 15. PMID 20156979
- [Result] Britto RR, Rezende NR, Marinho KC, Torres JL, Parreira VF, Teixeira-Salmela LF. Inspiratory muscular training in chronic stroke survivors: a randomized controlled trial. Arch Phys Med Rehabil. 2011 Feb;92(2):184-90. doi: 10.1016/j.apmr.2010.09.029. PMID 21272713
- [Derived] Parreiras de Menezes KK, Nascimento LR, Ada L, Avelino PR, Polese JC, Mota Alvarenga MT, Barbosa MH, Teixeira-Salmela LF. High-Intensity Respiratory Muscle Training Improves Strength and Dyspnea Poststroke: A Double-Blind Randomized Trial. Arch Phys Med Rehabil. 2019 Feb;100(2):205-212. doi: 10.1016/j.apmr.2018.09.115. Epub 2018 Oct 12. PMID 30316960